CLINICAL TRIAL: NCT00762567
Title: An Open-Label, Single-Dose Study Evaluating the Pharmacokinetics of Phenylephrine in Children and Adolescents
Brief Title: Phenylephrine Pediatric Pharmacokinetic Study
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Johnson & Johnson Consumer and Personal Products Worldwide (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: PHEALY1006
Record Dates: First submitted 2008-09-26; First posted 2008-09-30 (Estimated); Last update posted 2011-10-06 (Estimated); Status verified 2011-10

CONDITIONS: Rhinitis
MeSH Terms: conditions — Rhinitis | interventions — Oxymetazoline

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 1 (Experimental): phenylephrine
  Interventions: Drug: phenylephrine HCl

INTERVENTIONS:
Drug: phenylephrine HCl — A single dose of a liquid dosage form of phenylephrine HCl 2.5mg/5mL, using a weight-age dosing schedule
  Other Names: Children's Sudafed PE Nasal Decongestant Liquid

SUMMARY:
To characterize the pharmacokinetics of phenylephrine in two pediatric populations: children, ages 2 to <12 years, and adolescents, ages 12 to <18 years.

DETAILED DESCRIPTION:
This study has an open-label, single-dose classical pharmacokinetic design with no comparator treatment or group. At least twenty-four (24) children, ages 2 to <12 years, and twelve (12) adolescents, ages 12 to <18 years, with nasal symptoms due to hay fever or other upper respiratory allergies will complete the study. To ensure that younger children are represented, at least 35% (8) of the 24 children enrolled will range from 2 to <6 years of age.

ELIGIBILITY:
Inclusion Criteria:

* Male and female children and adolescents, ages 2 to < 18 years, with a minimum weight of 24 pounds will be eligible to participate. In addition, each subject will be > 5th percentile and < 95th percentile for weight based on age and gender.
* Subjects will have a body mass index (BMI) > 5th percentile and less than or equal to the 90th percentile for age and gender.
* Subjects who have a history of allergic rhinitis and who are experiencing nasal symptoms associated with hay fever or other upper respiratory allergies will be included.
* Subjects and parents or legally authorized representatives who, in the investigator's view, are likely to be compliant and complete the study will be eligible to participate.
* Post menarchal female subjects must have a negative urine pregnancy test at screening and at Visit 2 on Day 1 before study medication is administered.
* Post menarchal female subjects must have practiced abstinence or use an effective form of birth control (e.g., intrauterine device, oral contraceptives, contraceptive implants or injections, diaphragm with spermicide, cervical cap, or consort use of condom) for at least three months before being enrolled in the study.
* Parents or legally authorized representatives have signed and dated an IRB-approved consent form for the subject to participate in the study indicating that the subject (and/or a legally acceptable representative) has been informed of all pertinent aspects of the study.
* Subjects, ages 6 to < 18 years, who have provided written assent to participate in the study

Exclusion Criteria:

* Evidence or history of clinically significant hematological, renal, endocrine, pulmonary, gastrointestinal, cardiovascular, hepatic, psychiatric, or neurologic disease.
* Findings from the medical history or physical examination with vital sign measurements that are not within the range of clinical acceptability.
* Have a known sensitivity or allergy to phenylephrine or EMLA cream.
* Took any prescription or nonprescription medication (except vitamins and/or fluoride supplements) within seven days before the study's start date.
* Drank any fruit juices (i.e., apple, orange, or grapefruit) within two days prior to the study start.
* Use of any monoamine oxidase inhibitor within two weeks prior to the dose of phenylephrine.
* Participated in, or completed, another clinical trial within seven weeks before the study's start date.
* Have a history of drug, alcohol, and tobacco use (older children and adolescents).
* Have a history of hepatitis B, a previous positive test for hepatitis B surface antigen, or a previous positive hepatitis C antibody.
* Have a history of HIV infection or previous demonstration of HIV antibodies.
* Pregnant or nursing females; females of childbearing potential who are unwilling or unable to use an acceptable method of nonhormonal contraception from at least three months prior to the first dose of study medication until completion of follow-up procedures.
* Relationship to persons involved directly with the conduct of the study (ie, principal investigator; subinvestigators; study coordinators; other study personnel; employees or contractors of the sponsor or its subsidiaries; and the families of each).

Ages: 2 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 36 (Actual)
Dates: Start 2008-09; Primary Completion 2008-11 (Actual); Study Completion 2008-11 (Actual)

PRIMARY OUTCOMES:
Pharmacokinetic Parameters | 10, 20, 30, 45, and 60 minutes, and at 1.5, 2, 2.5, 3, and 3.5 hours after the dose. For children >6, an additional blood sample will be collected at 4.5 hours after dosing

SECONDARY OUTCOMES:
For children 5 years and older and adolescents, the total amount of phenylephrine and its metabolites excreted, percent of the administered dose will be estimated from the urine samples along with the formation clearance of each metabolite. | 24 hours
Safety Assessments will consist of monitoring and recording all non-serious Adverse Events (AEs) and Serious Adverse Events (SAEs), their frequency, severity, seriousness, and relationship to the investigational product. | throughout duration of the study + 2 days (+30 days for spontaneously reported SAEs)

CONTACTS AND LOCATIONS:
Overall Officials: Dolly Parasrampuria, PhD, Study Director — McNeil Consumer Healthcare Division of McNEIL-PPC, Inc.
Locations (1):
- West Coast Clinical Trials, Cypress, California, United States

REFERENCES:
- [Derived] Gelotte CK, Parasrampuria DA, Zimmerman BA. Single-Dose Pharmacokinetics and Metabolism of the Oral Decongestant Phenylephrine HCl in Children and Adolescents. Pulm Ther. 2023 Mar;9(1):139-150. doi: 10.1007/s41030-022-00206-8. Epub 2022 Dec 8. PMID 36480111